CLINICAL TRIAL: NCT04130841
Title: Effects of Internal Limiting Membrane Peeling on Visual Function in Epiretinal Membrane Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Un Chul Park, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1901-159-1006
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Retinal Disease; Epiretinal Membrane
Keywords: Internal limiting membrane peeling
MeSH Terms: conditions — Retinal Diseases; Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous ILM peeling (Experimental)
  Interventions: Procedure: Internal Limiting Membrane Peeling
- Active ILM peeling (Active Comparator)
  Interventions: Procedure: Internal Limiting Membrane Peeling
- No ILM peeling (No Intervention)

INTERVENTIONS:
Procedure: Internal Limiting Membrane Peeling — After removal of the epiretinal membrane, indocyanine green staining will be used to determine the internal limiting membrane (ILM) peeled off with the epiretinal membrane. (Group 1: spontaneous ILM peeling) If it is confirmed that the internal limiting membrane is not peeled together, the investigators determine whether the active Internal limiting membrane peeling is performed by 1:1 randomization immediately during surgery. (Group 2: Active ILM peeling, Group 3: no ILM peeling) The outcomes of the three groups will be compared.
  Arms: Active ILM peeling; Spontaneous ILM peeling

SUMMARY:
The patients who are diagnosed with idiopathic epiretinal membrane and scheduled to undergo epiretinal membrane removal will be treated with conventional vitrectomy and the epiretinal membrane will be removed. After removal of the epiretinal membrane, indocyanine green staining will be used to determine the internal limiting membrane (ILM) peeled off with the epiretinal membrane. (Group 1: spontaneous ILM peeling) If it is confirmed that the internal limiting membrane is not peeled together, the investigators determine whether the active Internal limiting membrane peeling is performed by 1:1 randomization immediately during surgery. (Group 2: Active ILM peeling, Group 3: no ILM peeling) The outcomes of the three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or older than 19 years
* Patients diagnosed with idiopathic epiretinal membrane and scheduled to undergo the epiretinal membrane removal surgery

Exclusion Criteria:

* Accompanied with retinal vascular disease or intraocular inflammation
* Prior treatment with vitrectomy in the study eye
* History of glaucoma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-09-29 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Epiretinal membrane recurrence | 12 months after the surgery
  Recurrence of the epiretinal membrane after the surgery

SECONDARY OUTCOMES:
Best-corrected visual acuity | 12 months after the surgery
M-chart | 12 months after the surgery
Aniseikonia | 12 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Un Chul Park, Principal Investigator — Associate Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No